CLINICAL TRIAL: NCT03055728
Title: Rapid Strep Testing in Children With Recent Streptococcal Pharyngitis
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0388
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Streptococcal Infections
Keywords: streptococcal infections; rapid strep testing; rapid antigen detection test
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Throat swabs of the posterior oropharynx will be tested for rapid antigen test and throat culture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 / Study Group: Subjects presenting with signs or symptoms of acute pharyngitis, with a history of culture-proven GAS infection and subsequent 10-day antibiotic treatment within the preceding 28 days. Subjects will have a rapid strep antigen detection test and a throat culture to determine presence of strep.
  Interventions: Diagnostic Test: Rapid strep antigen detection test; Diagnostic Test: throat culture
- Group 2 / Control Group: Subjects presenting with signs or symptoms of acute pharyngitis, without a recent history of GAS infection. Subjects will have a rapid strep antigen detection test and a throat culture to determine presence of strep.
  Interventions: Diagnostic Test: Rapid strep antigen detection test; Diagnostic Test: throat culture

INTERVENTIONS:
Diagnostic Test: Rapid strep antigen detection test — Pharyngeal swab for rapid antigen detection of streptococcus
  Other Names: rapid strep
Diagnostic Test: throat culture — Pharyngeal swab for culture for bacteria (specifically streptococcus) presence

SUMMARY:
The purpose of this study is to determine if the rapid antigen detection test for Group A streptococcal pharyngitis diagnosis might yield higher rates of false positive results in patients who have been treated for GAS pharyngitis within 28 days of the test.

DETAILED DESCRIPTION:
Strep pharyngitis, or strep throat, is a common infection afflicting children, aged 2 and above. Testing for strep pharyngitis consists of a rapid test and/or a throat culture. However, it has been observed that rapid testing may not be accurate in children with a recent history of strep pharyngitis. Therefore, this study aims to determine the accuracy of rapid strep testing in children who are presenting with symptoms of strep throat, who also have a recent history of and treatment for strep pharyngitis. By demonstrating an inaccuracy in rapid strep testing in patients with a recent history of strep pharyngitis, unnecessary testing and antibiotic use may be decreased, thereby reducing costs, overuse of antibiotics, and antibiotic resistance.

The participants in the study will include 600 children, aged 2 to 20 years old, selected from a private practice in Northern Virginia who present to the practice with signs or symptoms suggestive of acute pharyngitis. Subjects are children who are presenting with signs and symptoms suggestive of acute pharyngitis by the Centor criteria, including sore throat, fever, abdominal pain and cervical lymphadenitis. Any child with above presenting symptoms who is to undergo Streptococcus rapid antigen testing will be recruited to participate in the study.

A letter of consent will be provided to the parents and guardians of the involved child, stating that the study will be voluntary and confidential, and that all results will be kept in a safe environment.

Investigators will be testing the difference between two proportions, the false positive rate in previously treated compared to those not treated.

ELIGIBILITY:
Inclusion Criteria:

* 2-20 years old
* Current signs and symptoms suggestive of acute pharyngitis, including sore throat, fever, abdominal pain and cervical lymphadenitis.

Exclusion Criteria:

* Potential subjects who have been treated with less than 10 days of antibiotic therapy
* Patients who report non-compliance with previous antibiotic therapy
* Patients who have already been included in the study and children with evidence of GAS carrier status

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants in the study will include 600 children, aged 2 to 20 years old, selected from a private practice in Northern Virginia who present to the practice with signs or symptoms suggestive of acute pharyngitis.
  Potential subjects who have been treated with less than 10 days of antibiotic therapy, patients who report non-compliance with previous antibiotic therapy, patients who have already been included in the study and children with evidence of GAS carrier status will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-05-09 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Rate of false positives and false negatives in rapid antigen testing compared to throat culture | 48-72 hours
  The primary objective is to use rapid antigen test results to compare the sensitivity and specificity of rapid antigen testing in children with symptoms of pharyngitis with and without a recent history of Group A streptococcus pharyngitis.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Barakat, MD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Northern Virginia Pediatrics, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheeler RD, Houston MS, Radke S, Dale JC, Adamson SC. Accuracy of rapid strep testing in patients who have had recent streptococcal pharyngitis. J Am Board Fam Pract. 2002 Jul-Aug;15(4):261-5. PMID 12150457
- [Background] Edmonson MB, Farwell KR. Relationship between the clinical likelihood of group a streptococcal pharyngitis and the sensitivity of a rapid antigen-detection test in a pediatric practice. Pediatrics. 2005 Feb;115(2):280-5. doi: 10.1542/peds.2004-0907. PMID 15687433
- [Background] McIsaac WJ, White D, Tannenbaum D, Low DE. A clinical score to reduce unnecessary antibiotic use in patients with sore throat. CMAJ. 1998 Jan 13;158(1):75-83. PMID 9475915
- [Background] Llor C, Calvino O, Hernandez S, Crispi S, Perez-Bauer M, Fernandez Y, Martinez T, Gomez FF, Cots JM. Repetition of the rapid antigen test in initially negative supposed streptococcal pharyngitis is not necessary in adults. Int J Clin Pract. 2009 Sep;63(9):1340-4. doi: 10.1111/j.1742-1241.2009.02048.x. PMID 19691618
- [Background] Leung AK, Newman R, Kumar A, Davies HD. Rapid antigen detection testing in diagnosing group A beta-hemolytic streptococcal pharyngitis. Expert Rev Mol Diagn. 2006 Sep;6(5):761-6. doi: 10.1586/14737159.6.5.761. PMID 17009909